CLINICAL TRIAL: NCT04166396
Title: Non-pulmonary Contributors of Exercise Intolerance in Patients With Cystic Fibrosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HM20016707
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
Keywords: resveratrol; nicotinamide riboside; exercise intolerance
MeSH Terms: conditions — Cystic Fibrosis | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A: Cystic fibrosis (Experimental): Patients with CF will be randomly assigned to resveratrol or placebo.
  Interventions: Drug: Resveratrol; Dietary Supplement: Placebo
- A: Healthy Controls (Experimental): Healthy controls will be randomly assigned to resveratrol or placebo
  Interventions: Drug: Resveratrol; Dietary Supplement: Placebo
- B: Cystic Fibrosis (Experimental): Patients with CF will be randomly assigned to NR or placebo.
  Interventions: Drug: NR; Dietary Supplement: Placebo
- B: Healthy Controls (Experimental): Healthy controls will be randomly assigned to NR or placebo
  Interventions: Drug: NR; Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Resveratrol — 500 mg resveratrol, BID
  Arms: A: Cystic fibrosis; A: Healthy Controls
Drug: NR — 500 mg NR BID
  Arms: B: Cystic Fibrosis; B: Healthy Controls
Dietary Supplement: Placebo — Placebo

SUMMARY:
The purpose of this research study is to examine if the use of antioxidant supplements impacts exercise intolerance in people with CF.

DETAILED DESCRIPTION:
Exercise intolerance is a critical problem for people with cystic fibrosis (CF) able to predict hospitalization independent of lung function. Recent studies have suggested that certain supplements may help improving exercise intolerance.

ELIGIBILITY:
Inclusion Criteria:

CF

* Diagnosis of CF
* Men and women (> 18 yrs. old)
* FEV1 percent predicted > 40%
* Patients with or without CF related diabetes
* Resting oxygen saturation (room air) >90%
* Traditional CF-antioxidant medications
* Ability to perform reliable/reproducible PFTs
* Clinically stable for 4 weeks (no exacerbations or need for antibiotic antioxidant within 4 weeks of testing or major change in medical status)
* Pancreatic sufficient and pancreatic insufficient patients

Exclusion Criteria:

CF

* Children 17 years old and younger
* FEV1<40% predicted
* Resting O2 saturation <90%
* Clinical diagnosis of heart disease
* Clinical diagnosis of PAH
* Febrile illness within 4 weeks of a study visit
* Antioxidant for pulmonary exacerbation within 4 weeks of a study visit
* Currently smoking, pregnant or nursing
* Vasoactive medications (i.e. nitrates, beta-blockers, Viagra etc.)
* Patients with B. Cepacia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Sirtuin1 (Sirt1) | Change from baseline to up to 20 weeks
  Sirt1 will be assessed via a standard assay from samples taken from the participant's vein

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rodriguez Miguelez, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States